CLINICAL TRIAL: NCT03225209
Title: Medically Reproducing Bariatric Surgery
Acronym: MRB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Moahad S Dar (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry); Durham VA Medical Center (U.S. Federal Agency); East Carolina University (Other)
Responsible Party: Sponsor-Investigator, Moahad S Dar, Principal Investigator, East Carolina University
Organization: East Carolina University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02050
Record Dates: First submitted 2017-07-05; First posted 2017-07-21 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Roux-en-y gastric bypass; GLP-1; Liraglutide; OPTIFAST
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: "Proof of concept" study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- OPTIFAST (Experimental): Subjects meeting inclusion criteria will be receive OPTIFAST meal replacement (MR) in the following manner:
  WK1-WK12 (5 MR/DAY)
  WK13-14 (4 MR/DAY)
  WK 15 (3 MR/DAY)
  WK 16 (2 MR/DAY)
  WK 17-18 (1 MR/DAY)
  WK 19-24 (No MR)
  Interventions: Other: OPTIFAST

INTERVENTIONS:
Other: OPTIFAST — OPTIFAST meal replacement includes shakes, bars and soups. These meal replacements will completely replace the subject's diet for the first 12 weeks of the study (baseline-week 12) followed by a gradual transition back to prepared meals over 6 weeks (week 13-18). Attempt will be made to reduce or eliminate Lantus and Metformin as long as glycemic control is maintained.

SUMMARY:
Type 2 diabetes (DM2) is a chronic disease affecting 29 million Americans and a leading cause of blindness, kidney failure, and limb loss (Engelgau et al 2004). Roux-en-Y gastric bypass (RYGB) is the only intervention that leads to durable DM2 remission ~ 80% of the time (Mingrone et al 2012). Yet, it's broad application is limited by cost, invasiveness, and clinical inertia. Medically reproducing RYGB would extend the benefit of disease remission to the vast majority of DM2 patients using a cheaper, less invasive and more palatable treatment approach. Although all of the mechanisms mediating DM2 remission are not known, it is widely accepted that RYGB induces caloric restriction and enhances meal-stimulated release of a gut-peptide called glucagon-like-peptide-1 (GLP-1) both of which improve glycemic control in type 2 diabetes (Dar et al 2012; Jackness 2013). Caloric restriction can be achieved using OPTIFAST which is a commercially available medical weight loss program that has demonstrated the ability to decrease weight and improve glycemic control (Kirschner et al; 1998). Enhanced meal-stimulated GLP-1 release can be achieved using Liraglutide an FDA-approved once daily GLP-1 analogue that improves glycemic control and induces weight loss.

The investigators hypothesize that adding OPTIFAST (caloric restriction) in suboptimally controlled DM2 patients on Liraglutide (enhanced meal stimulated GLP-1 release), Metformin and Lantus insulin will medically reproduce RYGB and lead to DM2 remission, weight loss, decreased medication intensity and improved health related quality of life.

DETAILED DESCRIPTION:
This is a 24 week "proof of concept" study that will examine if adding "caloric restriction" (OPTIFAST) to "enhanced GLP-1 release" (Liraglutide) will lead to discontinuation of Lantus and Metformin. The primary outcome measure is change in glycemic control measured as hemoglobin A1C. Secondary outcome measures are change in weight, medication intensity and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 25-70 years
* BMI > 30
* diagnosis of type 2 diabetes
* weight stable for 3 months
* hemoglobin A1C >7% and <10%
* on Liraglutide
* on Metformin
* on Lantus
* interested in losing weight
* agreeable to regular visits per study protocol
* access to telephone and reliable transportation
* has a VAMC provider

Exclusion Criteria:

* age >70
* A1C <7% or >10%
* current use of prandial insulin
* current use of sulfonylurea or any other oral agent except for Metformin
* current sue of any other basal insulin except for Lantus
* pregnant
* breast feeding
* prior history of pancreatitis
* prior history of gastroparesis
* history of thyroid cancer/multiple endocrine neoplasia/thyroid nodules/medullary thyroid cancer
* history of gallstones
* history of hyperoxaluria or calcium oxalate nephrolithiasis
* AST/ALT > 2 times the upper limit of normal
* current or past history of liver disease
* history of Roux-en-Y gastric bypass or gastric sleeve or any other bariatric procedure
* type 1 diabetes
* any gastrointestinal disease causing malabsorption
* unwilling or unable to complete scheduled testing
* thiazolidinedione use within past 6 months
* any serious and/or unstable medical, psychiatric, or other condition(s) that prevents the patient from providing informed consent or complying with the study
* organ transplantation or those on immunosuppressants
* chronic anticoagulation
* recent myocardial infarction, unstable angina, stroke, coronary artery bypass or transient ischemia attacks in the past 6 months
* chronic prednisone use
* peptic ulcer disease in past 6 months
* acute gastrointestinal disorders
* hepatitis
* cirrhosis
* GFR < 50
* deep vein thrombosis in the past 6 months
* bone fractures in the past 6 months
* lithium use
* active malignancy
* substance abuse
* unstable psychiatric condition
* history of suicidal ideation
* enrolled in another research study related to diet and/or physical activity

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Change in Glycemic control | Change in HbA1c from baseline at week 12 and week 24 will be measured
  Hemoglobin A1C (HbA1C) will be used to assess glycemic control during the study

SECONDARY OUTCOMES:
Change in Weight | Change in weight in kilograms from baseline at week 12 and week 24 will be measured
  Weight in kilograms will be used to assess weight change during the study
Change in Medication intensity | Change in MES from baseline at week 12 and week 24 will be measured
  Medication effect score (MES) will be used to assess medication intensity during the study
Change in Health Related Quality of Life (HRQOL) | Change in PAID from baseline at week 12, and week 24 will be measured
  Problem Areas in Diabetes Scale (PAID) is a well-validated measure used in clinical trials regarding diabetes and is a sensitive and specific measure of HRQOL.
Change in Health Related Quality of Life | Change in EQ-5D-5L from baseline at week 12 and week 24 will be measured
  EQ-5D-5L is a highly sensitive 5-item health status measure with good performance in Veteran outpatients. It assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in Physical activity | Change in IPAQ from baseline at week 12 and week 24 will be measured
  International Physical Activity Questionnaire (IPAQ) is a well validated tool to assess daily physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Moahad Dar, MD, Principal Investigator — Dept of Veteran Affairs
Locations (1):
- Department of Veteran Affairs, Greenville Health Care Center, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Dar MS, Chapman WH 3rd, Pender JR, Drake AJ 3rd, O'Brien K, Tanenberg RJ, Dohm GL, Pories WJ. GLP-1 response to a mixed meal: what happens 10 years after Roux-en-Y gastric bypass (RYGB)? Obes Surg. 2012 Jul;22(7):1077-83. doi: 10.1007/s11695-012-0624-1. PMID 22419108
- [Background] Engelgau MM, Geiss LS, Saaddine JB, Boyle JP, Benjamin SM, Gregg EW, Tierney EF, Rios-Burrows N, Mokdad AH, Ford ES, Imperatore G, Narayan KM. The evolving diabetes burden in the United States. Ann Intern Med. 2004 Jun 1;140(11):945-50. doi: 10.7326/0003-4819-140-11-200406010-00035. PMID 15172919
- [Background] Jackness C, Karmally W, Febres G, Conwell IM, Ahmed L, Bessler M, McMahon DJ, Korner J. Very low-calorie diet mimics the early beneficial effect of Roux-en-Y gastric bypass on insulin sensitivity and beta-cell Function in type 2 diabetic patients. Diabetes. 2013 Sep;62(9):3027-32. doi: 10.2337/db12-1762. Epub 2013 Apr 22. PMID 23610060
- [Background] Kirschner MA, Schneider G, Ertel NH, Gorman J. An eight-year experience with a very-low-calorie formula diet for control of major obesity. Int J Obes. 1988;12(1):69-80. PMID 3360564
- [Background] Mingrone G, Panunzi S, De Gaetano A, Guidone C, Iaconelli A, Leccesi L, Nanni G, Pomp A, Castagneto M, Ghirlanda G, Rubino F. Bariatric surgery versus conventional medical therapy for type 2 diabetes. N Engl J Med. 2012 Apr 26;366(17):1577-85. doi: 10.1056/NEJMoa1200111. Epub 2012 Mar 26. PMID 22449317